CLINICAL TRIAL: NCT04727307
Title: Neoadjuvant Atezolizumab and Adjuvant Atezolizumab + Bevacizumab in Combination With Percutaneous Radiofrequency Ablation of Small HCC: a Multicenter Randomized Phase II Trial
Brief Title: Neoadjuvant Atezo, Adjuvant Atezo + Beva Combined With RF Ablation of Small HCC: a Multicenter Randomized Phase II Trial
Acronym: AB-LATE02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL20_0094; 2024-519113-59-00 (EU CTIS Number); 2020-000569-18 (EudraCT Number)
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Atezolizumab; Bevacizumab; Percutaneous radiofrequency; Ablation; Liver disease
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases | interventions — atezolizumab; Neoadjuvant Therapy; Catheter Ablation; Bevacizumab; Adjuvants, Pharmaceutic; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant Atezolizumab before radiofrequency ablation then adjuvant Atezolizumab + Bevacizumab (Experimental): Neoadjuvant atezolizumab and adjuvant atezolizumab + bevacizumab in combination with percutaneous radiofrequency ablation
  Interventions: Drug: Atezolizumab (neoadjuvant); Procedure: Percutaneous Radiofrequency; Drug: Bevacizumab (adjuvant); Drug: Atezolizumab (adjuvant)
- Percutaneous radiofrequency ablation (Active Comparator): Percutaneous radiofrequency ablation, standard treatment
  Interventions: Procedure: Percutaneous Radiofrequency

INTERVENTIONS:
Drug: Atezolizumab (neoadjuvant) — Atezolizumab 1200mg will be delivered as an IV infusion on Day 1 of each cycle (every 3 weeks) in neoadjuvant, for 2 cycles. The initial dose will be delivered over 60 (± 15) minutes and if tolerated subsequent infusions may be given over 30 (± 10) minutes.
  Other Names: Tecentriq
  Arms: Neoadjuvant Atezolizumab before radiofrequency ablation then adjuvant Atezolizumab + Bevacizumab
Procedure: Percutaneous Radiofrequency — Any RFA system (uni/multi-needle, monopolar or multi-bi-polar) is allowed. Microwave ablation or irreversible electroporation is not allowed.
Drug: Bevacizumab (adjuvant) — Bevacizumab 15 mg/kg will be delivered as an IV infusion on Day 1 of each 3 week cycle in adjuvant, for 15 cycles maximum. The initial dose will be delivered over 90 minutes (±15 minutes) and if tolerated subsequent infusions may be given over 60 (± 10) minutes then over 30 (± 10) minutes.
  Other Names: Avastin 400 mg in 16 ml Injection; Avastin 100 mg in 4 ml Injection
  Arms: Neoadjuvant Atezolizumab before radiofrequency ablation then adjuvant Atezolizumab + Bevacizumab
Drug: Atezolizumab (adjuvant) — Atezolizumab 1200 mg will be delivered as an IV infusion on Day 1 of each cycle (every 3 weeks) in adjuvant, for 15 cycles maximum. The dose will be delivered over 30 (± 10) minutes.
  Other Names: Tecentriq
  Arms: Neoadjuvant Atezolizumab before radiofrequency ablation then adjuvant Atezolizumab + Bevacizumab

SUMMARY:
Following the results of study IMbrave150, the combination Atezolizumab + Bevacizumab is a promising treatment option for patients with HCC.

In addition, the high intrahepatic distant recurrence rate and accumulating evidence for a metastatic mechanism encourages exploring adjuvant/neoadjuvant strategies targeting tumor growth and metastatic escape in the context of percutaneous thermal ablation for small HCC.

Local ablation of HCC is therefore an "ideal" setting for testing atezolizumab + bevacizumab in combination with ablation, with the aim of reducing the risk of recurrence.

DETAILED DESCRIPTION:
Liver cancer is the sixth most common cancer and the third leading cause of death from cancer worldwide (source: Globocan 2018). Hepatocellular carcinoma (HCC) represents 80-90% of liver cancers. Percutaneous thermal ablation (PTA) is a validated treatment option for very early and early stage HCC, together with surgical resection and liver transplantation (EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma, J Hepatol 2018). Due to its excellent tolerance, particularly in patients with portal hypertension or bearing comorbidities, it now represents in France nearly 70% of the first-line curative treatment of "in Milan" tumours. The risk of local tumor progression (LTP) is ≈10-20% in PTA series (Nault, J Hepatol 2018; N'Kontchou et al., Hepatology (Baltimore, Md) 2009). In addition, the long-term results of PTA are influenced by the high rate (up to 60-80% at 5 years) of intrahepatic distant recurrence (IDR) (Nault et al., J Hepatol 2018), as observed also after HCC surgical resection (EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma, J Hepatol 2018; Imamura et al., J Hepatol 2003). It is unknown whether early IDR (2-3 years after PTA of <3 cm HCC) is due to metastatic spread or de novo carcinogenesis.

Strong scientific rationale and emerging clinical data suggest that the combined vascular endothelial growth factor (VEGF) / Programmed death-ligand 1 (PD-L1) blockade may be clinically beneficial in a number of tumor types, including HCC. Therefore, local ablation in HCC is an " ideal " context to test Atezolizumab + Bevacizumab in combination with ablation. The investigators hypothesized that the combo of Atezolizumab + Bevacizumab and radiofrequency ablation could improve recurrence-free survival (RFS) at 2 years.

The aim of this randomized multicentre phase II trial is to compare RFS at 2 years in the experimental arm (Atezolizumab + Bevacizumab + RF ablation) versus the control arm (RF ablation) according to HCC modified response evaluation criteria in solid tumours (mRECIST). Thus the proposed use here of Atezolizumab as first neoadjuvant, then in combination with Bevacizumab as adjuvants, should theoretically, and hopefully, limit the radiofrequency ablation (RFA) pro-tumor effects. The RFS current rate value of 45% corresponding to the standard procedure of RFA alone (i.e. in the Active Comparator arm) should be increasing to at least 65% because of the addition of the biotherapy (i.e. in the Experimental arm). The patients' recruitment timeframe is set at 36 months and the patient's follow-up timeframe is 5 years. 202 patients are to be included, 101 per arm.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age
2. Diagnostic of HCC based on Imaging (EASL guidelines)
3. Patients with HCC eligible for ablation as assessed by multidisciplinary board:

   * All HCC nodules <3cm
   * 1-3 nodules of HCC
4. At least one uni-dimensional measurable lesion by magnetic resonance imaging (MRI) according to modified RECIST criteria
5. Liver function status Child-Pugh Class A
6. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory tests:

   * Hemoglobin > 8.5 g/dL
   * Absolute neutrophil count ≥ 1500/mm3
   * Platelet count ≥ 50,000/ mm3
   * Total bilirubin ≤ 2 mg/dL (ou ≤ 34 µmol/ L).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x upper limit of normal (ULN)
   * Serum creatinine ≤ 1.5 x ULN
   * Lipase ≤ 2 x ULN
   * Prothrombin time > 50%
   * Glomerular Filtration Rate (GFR) ≥ 35 mL/min/1.73 m2
8. Life expectancy ≥ 3 months
9. Women of childbearing potential and men must agree to use adequate contraception
10. Patients affiliated to a Social Security System

Exclusion Criteria:

1. Patients with contraindications to ablation or atezolizumab or bevacizumab
2. Patients with contraindication to contrast medium intravenous injection either gadolinium or iodinate
3. Patients with contraindication to MRI
4. Prior liver transplantation
5. Child-Pugh B or C
6. Patients with mixed histology (HCC and cholangiocarcinoma, namely hepatocholangiocarcinoma), if a biopsy is available
7. Current or recent (≤ 10 days prior to initiation of study treatment) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose. Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR < 1.5 x ULN and aPTT is within normal limits within 14 days prior to initiation of study treatment. For prophylactic use of anticoagulants or thrombolytic therapies, the approved dose as described by local label may be used.
8. Current or recent (≤10 days prior to initiation of study treatment) use of aspirin (> 325 mg/day) or treatment with clopidogrel, dipyramidole, ticlopidine, or cilostazol.
9. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

   1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
   2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

      * Rash must cover < 10% of body surface area.
      * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
      * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids.
10. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need forsystemic immunosuppressive medication during study treatment, with the following exceptions:

    * Patients who received acute, low-dose systemic immunosuppressant medication or a onetime pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor confirmation has been obtained.
    * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
11. Portal vein invasion, whatever its extent, shown on baseline imaging
12. Prior chemo-embolization or radio-embolization.
13. Patients with extra-hepatic metastases, either previously-treated or not. One lung nodule (<5mm) is allowed. Calcified lung micronodules as well as typical intra-pulmonary lymph nodes are allowed. Hepatic hilum lymph node < 10mm (short axis) is allowed.
14. Prior surgery of HCC with micro- or macro-vascular invasion demonstrated at pathology.
15. Prior systemic treatment for HCC, in particular agents targeting T-cell costimulation or checkpoint pathways (including those targeting PD-1, PD-L1 or PD-L2, cluster of differentiation 137 (CD137), or cytotoxic T-lymphocyte antigen (CTLA-4)).
16. Patients with uncontrolled HBV infection and viral load above 500 IU/mL.
17. Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding. Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrollment. Patients who have undergone an EGD within 6 months of prior to initiation of study treatment do not need to repeat the procedure
18. Past or concurrent history of neoplasm other than HCC, except for in-situ carcinoma of the cervix uteri and/or non-melanoma skin cancer and superficial bladder tumors. Any cancer curatively treated > 3 years prior to study entry is permitted
19. Known history or symptomatic meningeal tumors
20. Grade 3 (severe) hypertension ≥160 and/or ≥100 mmHG (systolic and diastolic, according to NCI-CTCAE v5.0)
21. Patients with phaeochromocytoma
22. Ongoing infection : Hepatitis B is allowed if no active replication is present (HBV replication below 500 IU/mL) or Hepatitis C is allowed if no antiviral treatment is required
23. Clinically significant bleeding NCI-CTCAE version 5.0 ≥ Grade 3 within 30 days before enrolment (transfusion indicated)
24. Arterial or venous thrombotic or embolic events such as cerebrovascular accident, deep vein thrombosis or pulmonary embolism within 6 months before enrolment
25. Any psychological, familial, sociological, geographical or illness or medical condition that could jeopardize the safety of the patient and/or his compliance with the study protocol and follow-up procedure
26. Known history of human immunodeficiency virus (HIV) infection
27. Seizure disorder requiring medication
28. Non-healing wound, ulcer or bone fracture
29. Breast feeding
30. Pregnancy
31. Legal incapacity (persons in custody or under guardianship)
32. Deprived of liberty Subject (by judicial or administrative decision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 2 years after randomization
  The primary outcome is to compare recurrence-free survival in patients treated by radiofrequency ablation versus neoadjuvant atezolizumab followed by radiofrequency ablation followed by adjuvant atezolizumab and bevacizumab.Recurrence is evaluated by the local investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Boris GUIU, MD, PhD, Study Director — University Hospital, Montpellier
Locations (19):
- France (19):
  - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - Hôpital Jean Verdier, Bondy
  - Hôpital Beaujon, Clichy
  - Centre Georges François Leclerc, Dijon
  - CHU Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHU de Lille, Lille
  - Hôpital Saint Joseph, Marseille
  - CHU de Montpellier, Montpellier
  - CHRU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHU Nîmes, Nîmes
  - Hôpital Cochin, Paris
  - CH Perpignan, Perpignan
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - Institut Gustave Roussy, Villejuif